CLINICAL TRIAL: NCT07158502
Title: Prevention of Infections Associated With Implantable Cardiac Devices
Brief Title: Antimicrobial Strategy for Device Implantation
Status: Not yet recruiting | Type: Observational
Sponsor: University of Calabria (Other)
Responsible Party: Principal Investigator, Antonio Curcio, Professor, University of Calabria
Other Study IDs: 195/2025
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: CIED-related Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TauroPace Cohort
  Interventions: Drug: TauroPace Cohort

INTERVENTIONS:
Drug: TauroPace Cohort — After sterile opening of the vial, the entire content of TauroPace™ will be poured into single-use sterile trays. Following skin incision, the surgical site will be irrigated with 5 mL of TauroPace™ solution.
  The leads, device generator, and fixation sutures will then be thoroughly wiped using sterile gauze soaked in the solution. Once the leads are connected to the generator, the entire system will be treated again with TauroPace™ before being inserted into the pocket.
  At the end of the procedure, the final surgical site will be irrigated once more with an additional 5 mL of TauroPace™ using a sterile syringe. A full 100 mL vial of the solution will be used for each patient, ensuring continuous antimicrobial coverage throughout the procedure.
  Excess solution will be gently removed prior to surgical wound closure.

SUMMARY:
Infections associated with cardiovascular implantable electronic devices (CIEDs) represent one of the major postoperative complications in interventional cardiology. These infections-including lead-related endocarditis, subcutaneous pocket infections, and sepsis-are characterized by high rates of morbidity, mortality, and healthcare costs. According to current epidemiological data, the incidence of CIED-related infections is estimated to be around 0.5-2% within the first 12 months and may rise to 5% over long-term follow-up. These infections are associated with a mortality rate of up to 34% and often require device explantation and prolonged antibiotic therapy.

TauroPace™ is an antimicrobial solution based on taurolidine, a broad-spectrum, non-antibiotic agent that acts by disrupting bacterial biofilms and preventing microbial colonization. Taurolidine has a favorable safety profile, does not induce antibiotic resistance, and is already approved in Europe as a CE-marked medical device (Directive 93/42/EEC). The application of TauroPace™ to the surface of CIEDs prior to implantation may significantly reduce the incidence of infections compared to the current standard, which consists of irrigating the device pocket with sterile saline solution.

The aim of this study is to rigorously and systematically evaluate the effectiveness of TauroPace™ compared to standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical indication for CIED implantation or generator replacement
* Signed informed consent to participate in the study

Exclusion Criteria:

* Known allergy to taurolidine or any of the excipients
* Severe immunodeficiency status (e.g., patients undergoing chemotherapy, with AIDS, or immunosuppressed following organ transplantation)
* Life expectancy < 12 months due to severe comorbidities (e.g., metastatic cancer, end-stage organ failure)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing implantation or generator replacement of cardiovascular implantable electronic devices (CIEDs). Participants will be consecutively enrolled during routine clinical activity over the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of CIEDs related infections | From enrollment to the end of 12 months
  To determine the incidence of infections related to cardiovascular implantable electronic devices (CIEDs) at 12 months in patients who received TauroPace™ during the implantation procedure.

SECONDARY OUTCOMES:
Safety Profile of TauroPace™ | From enrollment to 1 week after implantation
  To detect and describe any adverse events potentially related to the use of TauroPace

IPD SHARING:
Plan to Share IPD: No